CLINICAL TRIAL: NCT07343973
Title: Post-Market Study for the Evaluation of the Efficacy and Safety of the OpHLINE Ophthalmic Viscosurgical Device (OVD) in Cataract Surgery
Brief Title: Post-Market Study on the Safety and Effectiveness of the OpHLINE OVD in Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: i+Med S.Coop. (Industry)
Collaborators: Hospital Universitario Araba (Other); Hospital Universitario Basurto (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OpHLINE-PIC01-2020
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Cataract Surgery
Keywords: Hyaluronic acid; Ophtalmic viscosurgical device; Cataract surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OpHLINE® 1.4% (Experimental): Patients undergoing cataract surgery received the OpHLINE OVD with 1.4% sodium hyaluronate. This formulation is designed to maintain the anterior chamber space and protect corneal endothelial cells while offering easier removal due to its lower viscosity.
  Interventions: Device: Cataract Surgery by Phacoemulsification with Posterior Chamber Intraocular Lens Implantation (OpHLINE 1.4%)
- OpHLINE® 2% (Experimental): Patients in this group were treated with the OpHLINE OVD containing 2% sodium hyaluronate. This intermediate concentration aims to provide enhanced space stability during surgical phases while balancing protection and handling characteristics.
  Interventions: Device: Cataract Surgery by Phacoemulsification with Posterior Chamber Intraocular Lens Implantation (OpHLINE 2%)
- OpHLINE® 3% (Experimental): This group received the OpHLINE OVD with 3% sodium hyaluronate, the highest concentration tested. It is intended to maximize space maintenance and tissue protection during surgery, though it may require more effort for removal due to its higher viscosity.
  Interventions: Device: Cataract Surgery by Phacoemulsification with Posterior Chamber Intraocular Lens Implantation (OpHLINE 3%)

INTERVENTIONS:
Device: Cataract Surgery by Phacoemulsification with Posterior Chamber Intraocular Lens Implantation (OpHLINE 1.4%) — Eligible patients underwent cataract removal by phacoemulsification, followed by implantation of a posterior chamber intraocular lens (IOL) in a single eye.
  The surgical procedure included the following steps:
  Capsulorhexis: creation of a continuous circular opening in the anterior capsule of the lens.
  Hydrodissection: injection of fluid to separate the capsule from the cortex. Phacoemulsification: ultrasonic fragmentation and aspiration of the opacified lens through a micro-incision.
  IOL insertion: placement of the intraocular lens in the posterior chamber.
  OpHLINE 1.4% OVD was used as an adjunct during these phases to maintain the anterior chamber space and protect ocular tissues. After lens implantation, the viscoelastic device were aspirated according to standard surgical practice.
  Arms: OpHLINE® 1.4%
Device: Cataract Surgery by Phacoemulsification with Posterior Chamber Intraocular Lens Implantation (OpHLINE 2%) — Eligible patients underwent cataract removal by phacoemulsification, followed by implantation of a posterior chamber intraocular lens (IOL) in a single eye.
  The surgical procedure included the following steps:
  Capsulorhexis: creation of a continuous circular opening in the anterior capsule of the lens.
  Hydrodissection: injection of fluid to separate the capsule from the cortex. Phacoemulsification: ultrasonic fragmentation and aspiration of the opacified lens through a micro-incision.
  IOL insertion: placement of the intraocular lens in the posterior chamber.
  OpHLINE 2% OVD was used as an adjunct during these phases to maintain the anterior chamber space and protect ocular tissues. After lens implantation, the viscoelastic device were aspirated according to standard surgical practice.
  Arms: OpHLINE® 2%
Device: Cataract Surgery by Phacoemulsification with Posterior Chamber Intraocular Lens Implantation (OpHLINE 3%) — Eligible patients underwent cataract removal by phacoemulsification, followed by implantation of a posterior chamber intraocular lens (IOL) in a single eye.
  The surgical procedure included the following steps:
  Capsulorhexis: creation of a continuous circular opening in the anterior capsule of the lens.
  Hydrodissection: injection of fluid to separate the capsule from the cortex. Phacoemulsification: ultrasonic fragmentation and aspiration of the opacified lens through a micro-incision.
  IOL insertion: placement of the intraocular lens in the posterior chamber.
  OpHLINE 3% OVD was used as an adjunct during these phases to maintain the anterior chamber space and protect ocular tissues. After lens implantation, the viscoelastic device were aspirated according to standard surgical practice.
  Arms: OpHLINE® 3%

SUMMARY:
This post-market clinical study was designed to assess the safety and effectiveness of the OpHLINE Ophthalmic Viscosurgical Device (OVD) as an adjunct in cataract surgery. OpHLINE is a sterile, viscoelastic solution based on high-molecular-weight sodium hyaluronate, intended to maintain the anterior chamber space and protect corneal endothelial cells during phacoemulsification and intraocular lens (IOL) implantation.

The hypothesis is that OpHLINE, available in three concentrations (1.4%, 2%, and 3%), will provide optimal space maintenance throughout all surgical phases-capsulorhexis, hydrodissection, phacoemulsification, and IOL insertion-while ensuring ease of removal and minimizing postoperative complications. Specifically, the study expects the device to demonstrate high biocompatibility, effective protection of corneal endothelial cells, and a low incidence of adverse events, including intraocular pressure (IOP) spikes.

The objectives include confirming compliance with current clinical performance standards and collecting surgeons' feedback on handling and usability. This evaluation aims to strengthen real-world evidence supporting OpHLINE as a safe and reliable solution for cataract surgery, ensuring patient safety and surgical efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older scheduled for cataract extraction by phacoemulsification, followed by implantation of a posterior chamber intraocular lens (IOL) in a single eye (operative eye).
* The non-operative eye must be functional, as assessed by the investigator.

Exclusion Criteria:

* Ocular hypertension (IOP ≥ 22 mmHg).
* Corneal endothelial damage (cell count < 2000 cells/mm²).
* History of chronic or recurrent ocular inflammatory disease.
* Chronic or recurrent uveitis.
* Acute ocular disease.
* Internal or external ocular infection.
* Glaucoma or proliferative diabetic retinopathy.
* Previous ocular trauma before surgery.
* Congenital ocular anomalies or iris atrophy.
* Any other ocular pathology or physiological condition that could be worsened by cataract surgery.
* Previous ocular surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Ability to maintain anterior chamber space during cataract surgery. | 90 days
  This outcome evaluates whether the OpHLINE OVD can maintain a stable and adequate anterior chamber throughout all critical phases of cataract surgery: capsulorhexis, hydrodissection, phacoemulsification, and intraocular lens (IOL) insertion. Surgeons assessed this parameter using a structured questionnaire, classifying the chamber status into four categories: Complete chamber, Adequate working space, Shallow chamber, and Flat. A positive outcome is defined as achieving either a complete chamber or adequate working space in at least 70% of cases. This measure reflects the core functionality of the OVD in providing surgical safety and facilitating precise maneuvers.
Safety evaluation of OpHLINE during and after surgery | 90 days
  This measure involves systematic monitoring and documentation of any serious adverse events related to the device during the entire study period. SAEs include any event that could result in significant harm or require medical intervention. The target is an incidence rate of ≤1%, confirming that the device does not introduce unexpected risks beyond those inherent to cataract surgery.

SECONDARY OUTCOMES:
Assessment of removal difficulty after IOL implantation | 6 hours
  Surgeons classify removal as Easy, Normal, or Problematic. Adequate removal is defined as Easy or Normal in at least 70% of cases
Percentage of endothelial cell density loss | 90 days
  Endothelial cell density was measured using a non-contact specular microscope at baseline and at 90 days post-surgery. The goal is to determine the protective effect of the OVD on corneal tissue during surgery. A loss of ≤12% is considered optimal, as excessive cell loss can compromise corneal transparency and visual outcomes.
Incidence of IOP ≥30 mmHg during follow-up | 90 days
  IOP was measured at all scheduled visits to monitor postoperative pressure changes. The target is ≤13% incidence at 6 hours post-surgery and ≤6% at subsequent visits. Elevated IOP (>30 mmHg) can lead to optic nerve damage if not controlled, so this measure ensures the device does not contribute to clinically significant pressure spikes.
Frequency of non-serious adverse events during follow-up | 90 days
  This includes any minor complications or events that occur during or after surgery, such as mild inflammation or transient discomfort. The acceptable threshold is ≤30% across the study period, aligning with typical postoperative profiles for cataract surgery.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Basurto University Hospital, Bilbao, Bizkaia
  - Araba University Hospital, Vitoria-Gasteiz, Álava

IPD SHARING:
Plan to Share IPD: No